CLINICAL TRIAL: NCT02949791
Title: Effects of High Intra-abdominal Pressure on Tissue Diffusion and Pharmacokinetics of Cisplatin During HIPEC
Brief Title: HIPEC Using High Intra-abdominal Pressure
Acronym: HIPEC-IAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Principal Investigator, Shigeki Kusamura, Dr.Shigeki Kusamura, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIRC-2013-144445
Record Dates: First submitted 2016-10-07; First posted 2016-10-31 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Pseudomyxoma Peritonei; Colorectal Cancer
Keywords: cisplatin; HIPEC; Intra abdominal pressure; tissue drug concentration
MeSH Terms: conditions — Pseudomyxoma Peritonei; Colorectal Neoplasms | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Intra abdominal pressure HIPEC (Active Comparator): Cytoreductive surgery and HIPEC with low intra-abdominal pressure
  Interventions: Procedure: Cytoreductive surgery; Other: Low Intra abdominal pressure HIPEC
- High Intra abdominal pressure HIPEC (Experimental): Cytoreductive surgery and HIPEC with high intra-abdominal pressure
  Interventions: Procedure: Cytoreductive surgery; Other: High Intra abdominal pressure HIPEC

INTERVENTIONS:
Procedure: Cytoreductive surgery — Maximal surgical effort to obtain a minimal residual disease of less than 2.5 mm
  Other Names: Peritonectomy procedures
Other: Low Intra abdominal pressure HIPEC — Hyperthermic intraperitoneal chemotherapy using closed modality and intra abdominal pressure of 8-12 mmHg
  Arms: Low Intra abdominal pressure HIPEC
Other: High Intra abdominal pressure HIPEC — Hyperthermic intraperitoneal chemotherapy using closed modality and intra abdominal pressure of 18-22 mmHg
  Arms: High Intra abdominal pressure HIPEC

SUMMARY:
Cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) is a promising therapy for peritoneal carcinomatosis (PC) of various origins. Rather than the pharmacokinetic advantage, the uptake of chemotherapy by tumor tissue has been proposed as the best pharmacologic endpoint to assure the efficacy of HIPEC.

The primary endpoints of the present phase II randomized study are to test whether the increased intra abdominal pressure (IAP) during HIPEC could:

* enhance the penetration of cisplatin into the residual neoplastic and normal tissues;
* elicit changes on pharmacokinetic advantage of cisplatin.

Secondary endpoints are to evaluate the:

* impact of high IAP on intraoperatory hemodynamic and respiratory parameters;
* impact on short-term surgical outcomes (in hospital stay, morbidity, mortality).

Patients affected by PC from colorectal cancer or pseudomyxoma peritonei, submitted to complete cytoreduction (residual disease <2.5mm) would be eligible for the study. HIPEC will be performed using closed abdomen technique and cisplatin + mitomycin-C. Patients will be randomly assigned to HIPEC with low IAP (8-12 mmHg) or high IAP (18-22 mmHg). IAP will be measured using bladder catheter. High IAP will be obtained increasing the volume of perfusate.

Thirty-eight patients (19 in each study groups) will be enrolled in 30 months. The randomized groups will be stratified according to tumor type.

DETAILED DESCRIPTION:
Patients affected by peritoneal metastasis from colorectal cancer or pseudomyxoma peritonei, submitted to complete cytoreduction (residual disease <2.5mm) would be eligible for the study. Residual and resectable tumour nodules of 0.5 to 1.0 cm will be left behind after the cytoreduction and they will be collected at the end of HIPEC for the purpose of this study. HIPEC will be performed using closed abdomen technique and cisplatin (42mg/L of perfusate) + mitomycin-C (3.3mg/m2/L of perfusate) for 60 minutes, at 42.5°C. Patients will be randomly assigned to HIPEC with low IAP (8-12 mmHg) or high IAP (18-22 mmHg). IAP will be measured using bladder catheter. Patients of high IAP group will be strictly monitored during the perfusion regarding hemodynamic/respiratory parameters. During the HIPEC, perfusate and blood samples will be collected every 10 minutes. Additional samples of arterial blood will be collected at 70, 90,120,180 and 240 minutes. After the completion of HIPEC residual tumor tissues, normal peritoneum and muscular fascia will be sampled for determination of cisplatin concentration.

Blood samples will be immediately centrifuged to separate plasma. An aliquot of plasma will be stored at -30°C for total platinum determination. Another aliquot will be ultrafiltered by centrifugation through a membrane with a cut-off 5000 Da for ultrafilterable platinum determination. The ultrafiltrate will be stored at -30°C until analysis.

Perfusate samples will follow the same procedure of blood samples. Tissues samples will be stored at -80°C until analysis. Platinum determination will be performed using an Inductive Coupled Plasma Mass Spectrometry (ICP-MS) system by Thermo Scientific after preparing calibration curves with atomic platinum. Fluid samples simply dilute before ICP-MS examination while tissues will be desiccated, digested with a mixture of nitric acid and oxygen water, and evaporated to dryness prior to determination.

The investigators will compare the following outcomes between the study groups: tumor tissue concentration of cisplatin; the area under the curve (AUC) ratio of perfusate UF concentration of cisplatin times time to plasma UF concentration times time; in-hospital stay; systemic toxicity (NCI-CTCAE.v3), morbidity, and mortality.

Thirty eight patients (19 in each group) would be needed to detect an increase cisplatin concentration of 20 ng/mg of tumor tissue if patients are submitted to high-IAP during HIPEC, assuming alfa=0.05 and power=0.90 and standard deviation of 15 ng. Accrual time will be 30 months. The randomized groups will be stratified according to tumor type.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of primary peritoneal carcinomatosis from colorectal origin or pseudomyxoma peritonei
2. Patients submitted to complete cytoreduction with residual tumor <2.5 mm
3. Patients at the end of cytoreduction should present the laboratorial and hemodynamic parameters set as followings:

   * Mean arterial pressure > 65 mmHg
   * Heart rate: < 100 bpm
   * Central venous pressure > 4 mmHg
   * Cardiac index > 2.2
   * Central venous oxygen saturation (ScvO2) > 72%, and
   * Haemoglobin > 8.0 gr/dl.
4. Informed consent signed from the patient before the procedure.

Exclusion Criteria:

* Severe hemodynamic and/or respiratory instability after the cytoreduction that precludes HIPEC.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Tumor tissue concentration of cisplatin | collected within 15 minutes after the completion of HIPEC
  residual neoplastic tissue concentration of cisplatin measured in ng/mg
Normal tissue concentration of cisplatin | collected within 15 minutes after the completion of HIPEC
  tissue concentration of cisplatin measured in ng/mg in peritoneum of mesentery and rectal muscle fascia

SECONDARY OUTCOMES:
Pharmacokinetic advantage | During the HIPEC up to 1 hour from the completion of perfusion
  Peritoneal to plasma area under the curve (AUC) ratio of ultrafiltrated cisplatin concentrations
Pharmacokinetic advantage 2 | During the HIPEC up to 1 hour from the completion of perfusion
  Peritoneal to plasma area under the curve (AUC) ratio of total protein bound cisplatin concentrations
Impact of high intra-abdominal pressure on anesthesiologic parameters 1 | Intraoperative phase
  Mean arterial pressure (mmHg)
Impact of high intra-abdominal pressure on anesthesiologic parameters 2 | Intraoperative phase
  Heart rate (beats per minute)
Impact of high intra-abdominal pressure on anesthesiologic parameters 3 | Intraoperative phase
  Central venous pressure (mmHg)
Impact of high intra-abdominal pressure on anesthesiologic parameters 4 | Intraoperative phase
  Cardiac index
Impact of high intra-abdominal pressure on anesthesiologic parameters 5 | Intraoperative phase
  Arterial oxygen saturation (PaO2)
Impact of high intra-abdominal pressure on anesthesiologic parameters 6 | Intraoperative phase
  Central venous oxygen saturation (ScvO2)
Impact of intraoperative high intra-abdominal pressure on short-term surgical outcomes 1 | within 30 days after surgery
  Surgical complications (NCI CTCAEv3)
Impact of intraoperative high intra-abdominal pressure on short-term surgical outcomes 2 | within 30 days after surgery
  Systemic toxicity (NCI CTCAEv3)
Impact of intraoperative high intra-abdominal pressure on short-term surgical outcomes 3 | within 30 days after surgery
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Kusamura, MD PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esquis P, Consolo D, Magnin G, Pointaire P, Moretto P, Ynsa MD, Beltramo JL, Drogoul C, Simonet M, Benoit L, Rat P, Chauffert B. High intra-abdominal pressure enhances the penetration and antitumor effect of intraperitoneal cisplatin on experimental peritoneal carcinomatosis. Ann Surg. 2006 Jul;244(1):106-12. doi: 10.1097/01.sla.0000218089.61635.5f. PMID 16794395
- [Background] Facy O, Al Samman S, Magnin G, Ghiringhelli F, Ladoire S, Chauffert B, Rat P, Ortega-Deballon P. High pressure enhances the effect of hyperthermia in intraperitoneal chemotherapy with oxaliplatin: an experimental study. Ann Surg. 2012 Dec;256(6):1084-8. doi: 10.1097/SLA.0b013e3182582b38. PMID 22634898
- [Background] Facy O, Combier C, Poussier M, Magnin G, Ladoire S, Ghiringhelli F, Chauffert B, Rat P, Ortega-Deballon P. High pressure does not counterbalance the advantages of open techniques over closed techniques during heated intraperitoneal chemotherapy with oxaliplatin. Surgery. 2015 Jan;157(1):72-8. doi: 10.1016/j.surg.2014.06.006. Epub 2014 Jul 12. PMID 25027716
- [Background] Rossi CR, Foletto M, Mocellin S, Pilati P, De SM, Deraco M, Cavaliere F, Palatini P, Guasti F, Scalerta R, Lise M. Hyperthermic intraoperative intraperitoneal chemotherapy with cisplatin and doxorubicin in patients who undergo cytoreductive surgery for peritoneal carcinomatosis and sarcomatosis: phase I study. Cancer. 2002 Jan 15;94(2):492-9. doi: 10.1002/cncr.10176. PMID 11900234
- [Background] Jacquet P, Stuart OA, Chang D, Sugarbaker PH. Effects of intra-abdominal pressure on pharmacokinetics and tissue distribution of doxorubicin after intraperitoneal administration. Anticancer Drugs. 1996 Jul;7(5):596-603. doi: 10.1097/00001813-199607000-00016. PMID 8862729
- [Background] Van der Speeten K, Stuart OA, Sugarbaker PH. Pharmacokinetics and pharmacodynamics of perioperative cancer chemotherapy in peritoneal surface malignancy. Cancer J. 2009 May-Jun;15(3):216-24. doi: 10.1097/PPO.0b013e3181a58d95. PMID 19556908
- [Derived] Kusamura S, Azmi N, Fumagalli L, Baratti D, Guaglio M, Cavalleri A, Garrone G, Battaglia L, Barretta F, Deraco M. Phase II randomized study on tissue distribution and pharmacokinetics of cisplatin according to different levels of intra-abdominal pressure (IAP) during HIPEC (NCT02949791). Eur J Surg Oncol. 2021 Jan;47(1):82-88. doi: 10.1016/j.ejso.2019.06.022. Epub 2019 Jun 21. PMID 31262599